CLINICAL TRIAL: NCT06392477
Title: A Multicenter, Multiple Expansion Cohort Phase 1 Study Evaluating the Safety and Activity of SAR448501/DR-0201 as Multiple Ascending Doses in Patients With Relapsed/Refractory B Cell Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate the Safety and Activity of SAR448501/DR-0201 in Patients With Relapsed/ Refractory B-Cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DR-0201-ONC-001; DR0201ONC001 (Other: Sanofi Identifier); U1111-1328-7660 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAR448501 dose escalation (Experimental): SAR448501 will be administered for up to 52 weeks. Different cohorts with up to 8 dose levels will be included.
  Interventions: Drug: SAR448501

INTERVENTIONS:
Drug: SAR448501 — Bispecific antibody
  Other Names: DR-0201

SUMMARY:
This is an open-label, multiple ascending dose (MAD), phase 1 study in adult patients with relapsed or refractory (R/R) B cell non-Hodgkin lymphoma (B-NHL). The purpose of the study is to identify possible optimal biological dosage(s) by assessing safety, tolerability, pharmacokinetics (PK), pharmacodynamics, clinical activity and immunogenicity of SAR448501/DR-0201.

The study duration per participant will be approximately 3 years, including a screening period of up to 28 days, a treatment period of 52 weeks, a safety follow-up period of approximately 28 days and a long-term follow-up period of every 3 months until withdrawal of consent, participant death or study closure, whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

* Participants with R/R B-NHL which has failed at least 2 prior lines available life-prolonging standard therapy and without treatment options that are recognized to offer clinical benefit.
* Adequate marrow reserve, renal function, and hepatic function.
* Measurable disease defined as ≥ 1 bi-dimensionally measurable nodal lesion of > 1.5 cm in the longest dimension for participants with fluorodeoxyglucose (FDG)-avid disease for subtypes with nodular disease or at least one bi-dimensionally measurable extranodal lesion, defined as > 1.0 cm in its longest dimension.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Life expectancy of ≥ 12 weeks.
* Use of a highly effective contraceptive measure for all males and all females of childbearing potential during study through 180 days post last dose; Females of childbearing potential need to have a negative serum pregnancy test within 7 days prior to first dose.
* Tumor tissue block or 3 to 5 unstained slides from lymph node or other relevant biopsy collected in the past 12 months. Participants must be willing to provide a baseline and at least 1 on-treatment biopsy, unless not safely accessible.
* Participants who have received prior CAR-T therapy must be >60 days post CAR-T at day of first dosing.

Exclusion Criteria:

* Burkitt's or Burkitt's like lymphoma or lymphoplastic lymphoma.
* Current history of central nervous system (CNS) involvement by malignancy.
* Prior allogeneic stem cell transplantation except for those with follicular lymphoma (FL) and mantle cell lymphoma (MCL), who are excluded if transplant occurred less than 100 days prior to dosing or if they exhibit grade > 1 graft versus host disease.
* Prior solid organ transplantation.
* Autologous stem cell transplantation ≤ 100 days prior to dosing.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematous, rheumatoid arthritis, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjorgen's syndrome, Guillain-Barre-syndrome, multiple sclerosis vasculitis, or glomerulonephritis (participants with a remote history of, or well-controlled autoimmune disease, may be eligible).
* Major surgery in the last 28 days prior to dosing.
* Evidence of significant, uncontrolled concomitant disease that could affect compliance with study.
* Current or past history of CNS disease (participants with remote history of non-lymphoma CNS disease and with no residual neurologic deficits may be eligible to enroll).
* QT interval corrected by Fridericia's formula (QTcF) > 480 msec.
* Significant cardiovascular disease.
* Received any anticancer systemic therapy within 4 weeks prior to first drug administration or 5 half-lives of the drug, whatever is shorter. Treatment with corticosteroid ≤ 25 mg/day prednisone or equivalent is allowed. Inhaled and topical steroids are allowed.
* Known infection with HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Active infection at baseline requiring systemic treatment with antimicrobial, antifungal, or antiviral agents in the 2 weeks prior to dosing.
* Administration of a live, attenuated vaccine within 4 weeks prior to first drug administration or anticipation that such vaccine administration would be necessary during the course of the study.
* Another invasive malignancy in the last 2 years (except basal cell carcinoma or squamous cell carcinoma of the skin, asymptomatic prostate cancer requiring only hormonal therapy and with normal prostate-specific antigen for > 1 year, and tumors deemed by the investigator to be of low likelihood for recurrence).
* Prothrombin time/international normalized ratio (INR) and activated partial thromboplastin time or partial thromboplastin time (aPTT/PTT) > 1.3 × ULN or outside the therapeutic range of the local laboratory if receiving therapeutic anticoagulation that would affect the prothrombin time/INR, participants with a history of a hypercoagulation event within 6 months, or participants who have known hypercoagulation risk factors will be excluded.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2028-01-21 (Estimated); Study Completion 2028-02-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse event (TEAE) | Baseline to 28 days post last dose
Potential pharmacologically optimized dose/regimen(s) of SAR448501 / DR-0201 in participants with R/R B-NHL | Cycle 1 (Day 1 to Day 28)
  Potential pharmacologically optimized dose/regimen(s) of SAR448501/DR-0201 in participants with R/R B-NHL as determined using an integrated assessment of efficacy, safety, pharmacokinetic (PK)/pharmacodynamic (PD), and exposure-response relationships

SECONDARY OUTCOMES:
Response rate assessed for CLL | Baseline until disease progression (up to the end of treatment at Week 52)
  Response rate assessed for chronic lymphocytic leukemia (CLL) by International Workshop on Chronic Lymphocytic Leukemia (iwCLL). The iwCLL response is based on the overall physical examination and evaluation of blood and bone marrow: complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD).
Response rate assessed for all other B-NHL lymphomas | Baseline until disease progression (up to the end of treatment at Week 52)
  Response rate assessed for all other B-NHL lymphomas by Lugano response criteria. The Lugano response is based on the overall radiographic response: complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), not evaluable (NE) and not available (NA).
Duration of response/remission (DOR) | Baseline until disease progression (up to the end of treatment at Week 52)
  DOR is defined as the time between first disease response and date of disease progression or death due to any cause, whichever occurs first.
Complete response/remission rate (CRR) | Baseline until the end of treatment (Week 52)
  Proportion of participants who have a complete response/remission, based on the disease assessments by the Investigator.
Time to response (TTR in months) | Baseline until the end of treatment (Week 52)
  TRR is defined as the time between the first administration of investigational medicinal product (IMP) at Cycle 1 Day 1 (C1D1) until first documented disease response.
Progression-free survival (PFS) | Baseline until disease progression (up to the end of treatment at Week 52)
  PFS is defined as the time between the first administration of IMP at C1D1 and date of disease progression or death due to any case, whichever occurs first.
Overall survival (OS) | Baseline until disease progression (up to the end of treatment at Week 52)
  OS is defined as the time between the first administration of IMP (C1D1) and death due to any cause.
Assessment of pharmacokinetic (PK) parameters: AUC0-t | Baseline to 28 days post last dose
  Area under the plasma concentration versus time curve calculated using the trapezoidal method during a dosing interval (t)
Assessment of PK parameters: Cmax | Baseline to 28 days post last dose
  Maximum observed plasma concentration
Assessment of PK parameters: Tmax | Baseline to 28 days post last dose
  Time to reach Cmax
Assessment of PK parameters: terminal elimination half-life | Baseline to 28 days post last dose
  Time for the concentration to decrease in half
Incidence of anti-drug antibodies (ADAs) | Baseline to 28 days post last dose
  Incidence of anti-drug antibodies (ADAs) against SAR448501/DR-0201

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- Australia (5):
  - Investigational Site Number : 001-203, Camperdown, New South Wales
  - Investigational Site Number : 001-202, Townsville, Queensland
  - Investigational Site Number : 001-205, Adelaide, South Australia
  - Investigational Site Number : 001-204, Melbourne, Victoria
  - Investigational Site Number : 001-201, Perth, Western Australia
- Investigational Site Number : 001-703, Kamenitz, Serbia
- Singapore (2):
  - Investigational Site Number : 001-601, Singapore
  - Investigational Site Number : 001-602, Singapore
- South Korea (5):
  - Investigational Site Number : 001-401, Busan
  - Investigational Site Number : 001-403, Busan
  - Investigational Site Number : 001-404, Goyang-si
  - Investigational Site Number : 001-402, Seoul
  - Investigational Site Number : 001-405, Seoul
- Taiwan (3):
  - Investigational Site Number : 001-503, Changhua
  - Investigational Site Number : 001-502, Kaohsiung City
  - Investigational Site Number : 001-501, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org